CLINICAL TRIAL: NCT05376475
Title: Sleep in Late Pregnancy - Artificial Intelligence Development for the Detection of Disturbances and Disorders (SLeeP AID4): An Observational, In-Home, Single-Group, Feasibility Study
Brief Title: Sleep in Late Pregnancy - Artificial Intelligence Development for the Detection of Disturbances and Disorders
Acronym: SLeeP AID4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shiphrah Biomedical Inc. (Industry)
Collaborators: Mitacs (Industry); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: SBI-007
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy Related; Sleep; Sleep-Disordered Breathing; Sleep Disturbance; Sleep Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Virtual setup cohort: Participants in this cohort will use a night vision camera and level III home sleep apnea test. If the participant has a bed partner who consents to be in the study, the bed partner will also use a level III home sleep apnea test and be recorded by the night vision camera.
  Interventions: Device: Infrared video-audio camera; Device: Level III home sleep apnea test
- In-person setup cohort: Participants in this cohort will use a night vision camera, a level III home sleep apnea test, a maternal-fetal transabdominal electrocardiographic heart rate monitor, and a pressure sensing mat. If the participant has a bed partner who consents to be in the study, the bed partner will also use a level III home sleep apnea test and be recorded by the night vision camera (maternal-fetal transabdominal electrocardiographic heart rate monitor and a pressure sensing mat will not be used by the bed partner).
  Interventions: Device: Infrared video-audio camera; Device: Level III home sleep apnea test; Device: Maternal-fetal transabdominal electrocardiographic heart rate monitor; Device: Pressure sensing mat

INTERVENTIONS:
Device: Infrared video-audio camera — Wyze Cam V2 by Wyze Labs, Inc., Seattle, USA
Device: Level III home sleep apnea test — NightOwl® by Ectosense, Leuven, Belgium
Device: Maternal-fetal transabdominal electrocardiographic heart rate monitor — The Monica AN24 Antenatal Fetal Holter by Monica Healthcare, Nottingham, UK
  Groups: In-person setup cohort
Device: Pressure sensing mat — Tactilus® V Series Mattress Pressure Monitoring System by Sensor Products Inc., Madison, USA
  Groups: In-person setup cohort

SUMMARY:
SLeeP AID4 is a single-group, single-arm, Canada-wide, non-randomised, unblinded, in-home, observational study to prospectively collect and build a data set of natural sleep behaviour and physiology in maternal-fetal dyads (and bed partners, if applicable) in the third trimester of pregnancy in the home setting and subsequently investigate the feasibility of using computer vision technology (CVT) to monitor sleep during and across the third trimester of pregnancy in the home setting for research purposes by eliciting participants' attitudes toward CVT and training, validating, and testing a CVT model to accurately, unobtrusively, non-invasively, and objectively detect and quantify various sleep behaviours, disturbances, and disorders.

ELIGIBILITY:
Participant Inclusion Criteria:

* Healthy (see American Society of Anesthesiologists Physical Status [ASA-PS] classification; participant must be ASA-PS class II or lesser)
* Have a singleton pregnancy
* Be in the third trimester (gestational age between 28 weeks and 0 days through 40 weeks and 6 days, inclusive, by first-trimester ultrasound)
* Live in a home with a 2.4 GHz Wi-Fi network
* Sleep in a bed at night (i.e., not a La-Z-Boy chair or similar)

Participant's Bed Partner (if applicable) Inclusion Criteria:

* Sleep in the same bed as the pregnant study participant.
* Healthy (see American Society of Anesthesiologists Physical Status [ASA-PS] classification; participant must be ASA-PS class II or lesser)

Participant Exclusion Criteria:

* Non-English speaking, reading, or writing
* ASA-PS class III or greater

Participant's Bed Partner (if applicable) Exclusion Criteria:

* Non-English speaking, reading, or writing
* ASA-PS class III or greater

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant persons with singleton pregnancies in their third trimester living in Canada and their bed partner (if applicable).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal supine sleep position | 4 nights (approximately 32 hours)
  Average time per night, in minutes, spent supine while in bed as determined by manual review of infrared video.

SECONDARY OUTCOMES:
Bed partner sleep position | 4 nights (approximately 32 hours)
  Average time per night, in minutes, spent supine while in bed as determined by manual review of infrared video.
Maternal obstructive sleep apnea | 4 nights (approximately 32 hours)
  Average nightly Apnea-Hypopnea Index as determined by the home-sleep apnea test.
Bed partner obstructive sleep apnea | 4 nights (approximately 32 hours)
  Average nightly Apnea-Hypopnea Index as determined by the home-sleep apnea test.
Maternal limb movements | 4 nights (approximately 32 hours)
  Average nightly periodic limb movement index (number of limb movements per hour)
Bed partner limb movements | 4 nights (approximately 32 hours)
  Average nightly periodic limb movement index (number of limb movements per hour)
Maternal restless legs syndrome | 4 nights (approximately 32 hours)
  Present or absent, as determined by participant self report.
Bed partner restless legs syndrome | 4 nights (approximately 32 hours)
  Present or absent, as determined by participant self report.
Maternal total sleep time (TST) | 4 nights (approximately 32 hours)
  Average nightly total sleep time in minutes as determined by the home-sleep apnea monitor.
Bed partner total sleep time (TST) | 4 nights (approximately 32 hours)
  Average nightly total sleep time in minutes as determined by the home-sleep apnea monitor.
Maternal time in bed (TIB) | 4 nights (approximately 32 hours)
  Average nightly total time the participant is in bed.
Bed partner time in bed (TIB) | 4 nights (approximately 32 hours)
  Average nightly total time the participant is in bed.
Maternal sleep efficiency | 4 nights (approximately 32 hours)
  Average nightly percentage of total time in bed spent sleeping (ratio of TST to TIB multiplied by 100%).
Bed partner sleep efficiency | 4 nights (approximately 32 hours)
  Average nightly percentage of total time in bed spent sleeping (ratio of TST to TIB multiplied by 100%).
Maternal rapid eye movement (REM) sleep duration | 4 nights (approximately 32 hours)
  Average nightly time of REM sleep in minutes as determined by the home-sleep apnea monitor.
Bed partner rapid eye movement (REM) sleep duration | 4 nights (approximately 32 hours)
  Average nightly time of REM sleep in minutes as determined by the home-sleep apnea monitor.
Maternal snoring | 4 nights (approximately 32 hours)
  Present or absent as determined by manual review of audio from infrared video.
Bed partner snoring | 4 nights (approximately 32 hours)
  Present or absent as determined by manual review of audio from infrared video.
Minimum maternal heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly minimum HR, in beats per minute, as determined by the home-sleep apnea monitor.
Minimum maternal respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly minimum, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Minimum bed partner respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly minimum, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Minimum bed partner heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly minimum HR, in beats per minute, as determined by the home-sleep apnea monitor.
Minimum maternal peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly minimum, in percent, as determined by the home-sleep apnea monitor.
Minimum bed partner peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly minimum, in percent, as determined by the home-sleep apnea monitor.
Maximum maternal heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly maximum HR, in beats per minute, as determined by the home-sleep apnea monitor.
Maximum bed partner heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly maximum HR, in beats per minute, as determined by the home-sleep apnea monitor.
Maximum maternal respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly maximum, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Maximum bed partner respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly maximum, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Maximum maternal peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly maximum, in percent, as determined by the home-sleep apnea monitor.
Maximum bed partner peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly maximum, in percent, as determined by the home-sleep apnea monitor.
Average maternal heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly mean HR, in beats per minute, as determined by the home-sleep apnea monitor.
Average bed partner heart rate (HR) | 4 nights (approximately 32 hours)
  Averaged nightly mean HR, in beats per minute, as determined by the home-sleep apnea monitor.
Average maternal respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly mean, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Average bed partner respiration rate (RR) | 4 nights (approximately 32 hours)
  Averaged nightly mean, in breaths per minute, as determined by manual review of audio and video from the infrared video data.
Average maternal peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly mean, in percent, as determined by the home-sleep apnea monitor.
Average bed partner peripheral blood oxygen saturation (SpO2) | 4 nights (approximately 32 hours)
  Averaged nightly mean, in percent, as determined by the home-sleep apnea monitor.
Maternal heart rate variability - root mean square of successive differences | 4 nights (approximately 32 hours)
  Averaged nightly beat-to-beat variation as measured by the root mean square of successive differences (RMSSD).
Fetal heart rate variability - root mean square of successive differences | 4 nights (approximately 32 hours)
  Averaged nightly beat-to-beat variation as measured by the root mean square of successive differences (RMSSD).
Maternal heart rate variability - standard deviation of NN intervals | 4 nights (approximately 32 hours)
  Averaged nightly beat-to-beat variation as measured by the standard deviation of N-N intervals (SDNN).
Fetal heart rate variability - standard deviation of NN intervals | 4 nights (approximately 32 hours)
  Averaged nightly beat-to-beat variation as measured by the standard deviation of N-N intervals (SDNN).
Maternal skin pressure distribution thorax | 4 nights (approximately 32 hours)
  Averaged nightly mean pressure, in pounds per square inch (PSI), in the thorax region.
Maternal skin pressure distribution abdomen | 4 nights (approximately 32 hours)
  Averaged nightly mean pressure, in pounds per square inch (PSI), in the abdominal region.
Maternal skin pressure distribution pelvis | 4 nights (approximately 32 hours)
  Averaged nightly mean pressure, in pounds per square inch (PSI), in the pelvic region.
Average fetal heart rate (FHR) | 4 nights (approximately 32 hours)
  Averaged nightly mean FHR, in beats per minute, as determined by the ambulatory maternal-fetal heart rate monitor.
Minimum fetal heart rate (FHR) | 4 nights (approximately 32 hours)
  Averaged nightly minimum FHR, in beats per minute, as determined by the ambulatory maternal-fetal heart rate monitor.
Maximum fetal heart rate (FHR) | 4 nights (approximately 32 hours)
  Averaged nightly maximum FHR, in beats per minute, as determined by the ambulatory maternal-fetal heart rate monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Dolatabadi, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participants' study data will not be released outside of the study team without the written permission of the participant, except as necessary for duty to report or force of law (i.e., by subpoena). Study data will not be made open access.